CLINICAL TRIAL: NCT05301712
Title: A Placebo Controlled, Double-blind, Randomized, Multicenter Study to Evaluate the Efficacy and Safety of Naloxone HCl IV in Patients With Stroke
Brief Title: A Phase 4 Clinical Study to Investigate the Efficacy and Safety of Naloxone HCI IV in Patients With Stroke
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samjin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SJNLX01
Record Dates: First submitted 2022-03-11; First posted 2022-03-31 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Stroke, Acute
Keywords: cerebral infarction or cerebral hemmorrhage
MeSH Terms: conditions — Stroke; Cerebral Infarction | interventions — Naloxone; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This clinical trial was planned for the purpose of re-evaluating ischemic cerebral nerve disorders caused by stroke and cerebral hemorrhage the efficacy and effects of naloxone hydrochloride.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naloxone hydrochloride 5.0mg/5ml (Experimental): Naloxone hydrochloride 60mg (However, the dose may be appropriately increased or decreased according to the judgement of the investigator)
  Interventions: Drug: Naloxone hydrochloride 5.0mg/5ml
- Placebo (Placebo Comparator): Placebo 60ml (However, the dose may be appropriately increased or decreased according to the judgement of the investigator)
  Interventions: Drug: Sodium Chloride 45mg/5ml

INTERVENTIONS:
Drug: Naloxone hydrochloride 5.0mg/5ml — * Initial dose: 4mg, Intravenous injection
  * Continuous dose: 8mg(mixed with 1000ml of 5% Dextrose water or saline solution) per day, Intravenous infusion for 7days
  * Total dose: 4mg+8mg/day*7=60mg
  Other Names: Noloxone hydrochloride 5mg
  Arms: Naloxone hydrochloride 5.0mg/5ml
Drug: Sodium Chloride 45mg/5ml — * Initial dose: 4ml, Intravenous injection
  * Continuous dose: 8ml (mixed with 1000ml of 5% Dextrose water or saline solution) per day, Intravenous infusion for 7days
  * Total dose: 4ml+8ml/day*7=60ml
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This clinical trial was planned for the purpose to re-evaluate the safety and efficacy of naloxone hydrochloride in ischemic cerebral nerve disorders caused by stroke and cerebral hemorrhage.

Eligible subjects will be randomized to the naloxone hydrochloride group or placebo group at 1:1 ratio.

Also, factors, such as disease subtype and severity, which might impact the efficacy endpoints will be used to stratify.

- Stratification factor: cerebral infarction (NIHSS 5-15 points or 16-20 points) or cerebral hemorrhage

Administration of investigational product should be started within 48 hours from the onset of symptoms.

Subject receive the investigational product 7 consecutive times (for 7 days) in a single dose of intravenous infusion for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are males or females aged ≥19 years
* Patients with a stroke who can administer drugs for clinical trials within 48 hours from stroke onset
* Patients with a NIHSS score of 5-20 or GCS score of 8-13 at screening assessment (In the case of cerebral infarction, the NIHSS is evaluated, and cerebral hemorrhage, the GCS is evaluated.)
* Patients with a mRS(Modified Rankin Score) > 2 after stroke and immediately before randomization.
* Patients who or whose representative voluntarily agrees to this study and has given a written informed consent.

Exclusion Criteria:

* Subjects with medical history of hypersensitivity reaction to investigational product or ingredients.
* Patients with non-narcotic central nerve inhibitors such as barbital drugs or respiratory depression caused by pathological causes.
* Patients who have not passed the wash-out time after administration of opioid analgesics.
* Subjects with Renal dysfunction whose creatine level is more than twice the normal upper limit in screening tests
* Subjects with Liver dysfunction whose AST/ALT level is more than three times the normal upper limit in screening tests.
* Subjects with Systolic blood pressure less than 90 mmHg or more than 220 mmHg during screening.
* Patients with a mRS > 2 before stroke onset.
* Patients with a history of epilepsy.
* Patients with myocardial infarction within 1 month.
* Pregnant or lactating women
* Patients who have passed more than 48 hours since the onset of symptoms.
* Subjects who received other therapeutic investigational product within the last 30 days.
* Patients who transient ischemic attack.
* Patients whose life expectancy is less than 3 months due to comorbidities other than stroke
* Thrombolysis (including non-drug treatments such as thrombolytic drugs and mechanical procedures used in thrombolysis) or extraventricular drainage (surgical treatment) has been performed or is scheduled to be performed.
* Thrombolytic agent used in thrombolysis[ex. Streptokinase, Alteplase, Anistreplase, Urokinase, Reteplase, Tenecteplase, Tissue-plasminogen activator (t-PA), Single-chain urokinase-type plasminogen activator (Scu-PA), Lanoteplase, Monteplase, Plasminogen activator inhibitors (PAI)]
* Surgical treatment [ex. mechanical thrombectomy, external ventricular drainage (EVD), extralesional drainage (ELD), decompression], Subarachnoid hemorrhage (SH), Trauma patients [ex. SH coiling, traumatic intracranial hemorrhage (ICH)], Among patients with infarction, patients who need or are scheduled to perform Depressive craniomy.
* Any condition that, in the opinion of the investigator, would inappropriate to participate in the clinical trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects who have the modified Rankin Scale (mRS) score of 2 or less on Day 90 | Day 90
  Modified Rankin Scale is an index that evaluates the patient's global functional outcome according to the independence of daily life and the degree of need for help from others. It is evaluated in seven stages (0 to 6 points), from asymptomatic to death. The higher score means a worse outcome, and 3 to 6 points are considered to be poor functional outcome.

SECONDARY OUTCOMES:
The change from baseline in Modified Rankin Score (mRS) up to Day 90 | Baseline, Day 3, Day 7, Day 14(or discharge), Day 30 and Day 90
  Modified Rankin Scale is an index that evaluates the patient's global functional outcome according to the independence of daily life and the degree of need for help from others. It is evaluated in seven stages (0 to 6 points), from asymptomatic to death. The higher score means a worse outcome, and 3 to 6 points are considered to be poor functional outcome.
The change from baseline in Modified Barthel Index (mBI) up to Day 90. | Baseline, Day 3, Day 7, Day 14(or discharge), Day 30 and Day 90
The change from baseline in EuroQol five dimensions questionnaire(EQ-5D) up to Day 90 | Baseline, Day 3, Day 7, Day 14(or discharge), Day 30 and Day 90
The change from baseline in Korean Mini-Mental State Examination(KMMSE) up to Day 90 | Baseline, Day 3, Day 7, Day 14(or discharge), Day 30 and Day 90
The change from baseline in Global Deterioration Scale (GDS) up to Day 90 | Baseline, Day 3, Day 7, Day 14(or discharge), Day 30 and Day 90
  The GDS is a staging scale indicating deterioration in dementia, The scale details clinical descriptions of seven major distinguishable stages, ranging from normal cognition to severe dementia.
  Stages 1 - 3 are the pre dementia stages. Stages 4 -7 reflect the stages of dementia. People beginning with stage 5 are no longer survive without assistance.
The change from baseline in National institutes of health stroke scale(NIHSS) up to Day 90 | Baseline, Day 3, Day 7, Day 14(or discharge), Day 30 and Day 90
  It will be evaluated in patients with cerebral infarction.
  The NIHSS is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke.
  The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4.
  For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment.
  The individual scores from each item are summed in order to calculate a patient's total NIHSS score.
  The maximum possible score is 42, with the minimum score being a 0.
The change from baseline in Glasgow Coma Scale(GCS) up to Day 90 | Baseline, Day 3, Day 7, Day 14(or discharge), Day 30 and Day 90
  It will be evaluated in patients with cerebral hemorrhage. The Glasgow Coma Scale (GCS) is used to objectively describe the extent of impaired consciousness in all types of acute medical and trauma patients.
  The Glasgow Coma Scale divides into three parameters: best eye response (E), best verbal response (V) and best motor response (M). The levels of response in the components of the Glasgow Coma Scale are 'scored' from 1, for no response, up to normal values of 4 (Eye-opening response) 5 ( Verbal response) and 6 (Motor response) The total Coma Score thus has values between three and 15, three being the worst and 15 being the highest.
The odds ratio of the factors which contribute to a mRS score to be less than or equal to 2 on Day 90 | Day 90
  The factors, such as sex, age, disease subtype and severity, investigational product compliance, which might impact the mRS score to be less than or equal to 2 will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Keun Hyun, M.D.,Ph.D, Principal Investigator — Inha University Hospital
Locations (1):
- Inha University Hospital, Incheon, South Korea